CLINICAL TRIAL: NCT05751655
Title: Observational Study of Drowning Patient's Emergency Care in Its Pre-hospital Phase.
Acronym: VAR-NOYADE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-CHITS-002
Record Dates: First submitted 2023-02-10; First posted 2023-03-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Drowning
Keywords: Drowning; Emergency medical service; Pre-hospital care; Patient outcome
MeSH Terms: conditions — Drowning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Drowning patients: Process of experiencing respiratory impairment from submersion/immersion in liquid
  Interventions: Other: Prehospital care following drowning accident

INTERVENTIONS:
Other: Prehospital care following drowning accident — Prehospital care provided by the emergency medical service 83 (SAMU 83)

SUMMARY:
According to the 9th edition of "NOYADES" survey, 1480 drownings accidents occurred in France in 2021, of which 146 (i.e. nearly 10%), were in the Var department. These patient's care involve in first place the Emergency Medical Service (EMS).

To date, there is no recommendation from French or European academic societies of emergency medicine formalising pre-hospital care of these patients (except for the specific case of cardiac arrest). This absence of recommendation therefore favours heterogeneity of practices.

DETAILED DESCRIPTION:
Within a three-year period from 2019 to 2022, this retrospective observational study aims to provide an inventory of pre-hospital practices by the EMS in the Var department and to describe drowning patients' characteristics as well as their outcome, according to the initial regulation and the type of care. These data could help for pre-hospital care management.

ELIGIBILITY:
Inclusion Criteria:

1. Drowning patient
2. Aged 18 years old or over
3. Patient treated by pre-hospital care from the emergency medical services 83 (SAMU 83) between 1st January 2019 and 30th September 2022.

Exclusion Criteria:

1. Diving accident
2. Patient opposition to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult drowning patient treated by pre-hospital care from the emergency medical services 83 (SAMU 83) between 1st January 2019 and 30th September 2022.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Type of ventilation used in pre-hospital care | 3-year period from 2019-2022
  Mechanical ventilation, non-invasive ventilation, Continuous Positive Airway Pressure, oxygen therapy or none
Ventilatory settings used in pre-hospital care | 3-year period from 2019-2022
  Positive End Expiratory Pressure, pressure support, fraction of inspired oxygen, flow rate
Pre-hospital intervention duration | 3-year period from 2019-2022
  In minutes
Type of resources involved for pre-hospital care | 3-year period from 2019-2022
  None, fire brigade or emergency rapid response unit

SECONDARY OUTCOMES:
Onset of death | Up to 30 days
  Analysis according to the orientation provided by the EMS regulation (emergency rapid response unit or fire brigade) and according to the different types of care by the EMS (Oxygen therapy, non-invasive ventilation or intubation).
Duration of hospitalisation | Up to 30 days
  Analysis according to the orientation provided by the EMS regulation (emergency rapid response unit or fire brigade) and according to the different types of care by the EMS (Oxygen therapy, non-invasive ventilation or intubation).
Intubation rate at hospital | Up to 30 days
  Analysis according to the orientation provided by the EMS regulation (emergency rapid response unit or fire brigade) and according to the different types of care by the EMS (Oxygen therapy, non-invasive ventilation or intubation).
Type of ventilation used at hospital | Up to 30 days
  Analysis according to the orientation provided by the EMS regulation (emergency rapid response unit or fire brigade) and according to the different types of care by the EMS (Oxygen therapy, non-invasive ventilation or intubation).

CONTACTS AND LOCATIONS:
Overall Officials: Célia BOUTIN, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mathais Q, Jurain L, Sebai A, Mattei P, Jammes D, Kaidomar M, Kleiner G, Rammal F, Marquer B, Bertrand PM, Belloni A, Benner P, Meaudre E, Vergne M, Chelly J, Boutin C. Prehospital factors associated with ICU admission in drowning patients: a retrospective multicenter cohort study in a French coastal region. BMC Emerg Med. 2026 Jan 20. doi: 10.1186/s12873-026-01481-3. Online ahead of print. No abstract available. PMID 41559630